CLINICAL TRIAL: NCT03354039
Title: Tamoxifen in Duchenne Muscular Dystrophy: A Multicenter, Randomised, Double-blind, Placebo-controlled, Phase 3 Safety and Efficacy 48-week Trial
Brief Title: Tamoxifen in Duchenne Muscular Dystrophy
Acronym: TAMDMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAMDMD
Record Dates: First submitted 2017-10-10; First posted 2017-11-27 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamoxifen 20 mg once daily (Experimental): DMD patients randomised to verum will receive 20 mg (0.6mg/kg) of TAM daily.
  Interventions: Drug: Tamoxifen
- Matching placebo once daily (Placebo Comparator): Patients randomised to placebo will be administered matching placebo.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Tamoxifen — DMD patients randomised to verum will receive 20 mg (0.6mg/kg) of Tamoxifen daily. Treatment will be given for the total period of 48 weeks.
  Arms: Tamoxifen 20 mg once daily
Drug: Matching placebo — Patients randomised to placebo will be administered matching placebo. Treatment will be given for the total period of 48 weeks.
  Arms: Matching placebo once daily

SUMMARY:
A randomised, double blind, placebo controlled, 48-week clinical trial with a core population (group A) of 79 ambulant 6.5 to 12 years old Duchenne's muscular dystrophy (DMD) patients that are under stable standard treatment of care with glucocorticoids. Furthermore, the investigators plan to include 6-20 non-ambulant patients who do not receive glucocorticoids (as parallel group B), 10 to 16 years old, to obtain efficacy and safety data in a broader DMD population. All patients will receive 20 mg of tamoxifen (TAM) or placebo once daily during 48 weeks.

An open label extension (OLE) trial for participants of the TAMDMD main study will be performed. All TAMDMD patients on TAM or placebo are offered to enter this OLE.

DETAILED DESCRIPTION:
This is a 48-week multicentre, parallel, randomised, double-blind, placebo controlled phase 3 safety and efficacy trial. There are two treatment arms: Tamoxifen (verum) and placebo (control), with treatment allocation of 1:1.

The investigators plan to screen at least 79 and to enroll at least 71 ambulant DMD patients aged between 6.5 and 12 years (group A) and 6 - 20 non-ambulant DMD patients aged between 10 and 16 years (group B). In order to reach statistical power, 60 ambulant patients (group A) need to complete the trial. Treatment with 20 mg Tamoxifen once daily will be given for the total trial duration of 48 weeks.

Only patients with glucocorticoids (standard treatment of care) will be included in group A (ambulant patients) and only non-glucocorticoid users in group B. At baseline as well as at the end of the study clinical, laboratory, and MRI measurements will be performed. These include the Motor Function Measure (MFM) scale, timed function tests, the 6 minute walking distance, quantitative muscle testing (QMT) and quantitative thigh muscle MRI, questionnaires. A physical examination, an ECG, vital signs as well as safety laboratory blood analyses will be performed at every visit. Furthermore, an x-ray of the hand and a dual energy x-ray absorptiometry (DEXA)-scan will be performed at baseline and at the end of the study.

An open label extension (OLE) trial for participants of the TAMDMD main study will be performed. All TAMDMD patients on TAM or placebo are offered to enter this OLE. All OLE patients will receive 20 mg of TAM daily during 48 weeks. The same study specific assessments as in the double-blind randomized phase will be performed during the OLE phase

ELIGIBILITY:
Inclusion Criteria:

Group A (ambulant patients)

* Documented diagnosis of DMD by mutation analysis in the dystrophin gene or by substantially reduced levels of dystrophin protein (i.e. absent or <5% of normal) on Western blot or immunostaining
* Stable treatment with glucocorticoids >6 months (no significant change in dosage (>0.2mg/kg)) at screening; dosing adaptations according to weight change are allowed
* Male gender
* 6.5 to 12 years of age at time of screening
* weight >20kg
* ambulant patients
* able to walk at least 350 meters in 6 minute walking distance test without assistance at screening
* MFM D1 subdomain of the MFM scale >40% at screening
* Ability to provide informed consent and to comply with study requirements
* Patients harbouring a nonsense mutation treatable with the approved drug ataluren should be under stable ataluren treatment for at least 3 months or in case of nontolerance being off ataluren treatment for at least 3 months before screening

Group B (non-ambulant patients)

* Documented diagnosis of DMD by mutation analysis in the dystrophin gene or by substantially reduced levels of dystrophin protein (i.e. absent or <5% of normal) on Western blot or immunostaining
* Not using glucocorticoids for >6 months
* Male gender
* Non-ambulant patients (walking distance less than 10 meters)
* 10 to 16 years of age at time of screening
* Ability to provide informed consent and to comply with study requirements

Open label extension

- Recent participation and completion of TAMDMD study

Exclusion Criteria:

* Known individual hypersensitivity or allergy to tamoxifen or other ingredients/excipients of IMP
* Female gender
* Use of tamoxifen or testosterone within the last 3 months
* Known or suspected malignancy
* Other chronic disease or clinically relevant limitation of renal, liver or heart function
* Known or suspected non-compliance
* Any injury which may impact functional testing, e.g. upper or lower limb fracture
* Planned or expected spinal fusion surgery during the study period (as judged by the Investigator; i.e. due to rapid progressing scoliosis), previous spinal fusion surgery is allowed if it took place more than 6 months prior to screening.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders of the participant/parents (as judged by the investigator)
* Concomitant participation in any other interventional trial (and up to 3 months prior to screening)
* Use of CYP2D6 inhibitors or of CYP3A4 inducers (apart from glucocorticoids), platelet aggregation inhibitors and coumarin-type anti-coagulants
* Use of drugs metabolized by CYP2C9, such as phenprocoumon, phenytoin, warfarin, celecoxib, fluvastatin, ginko biloba, St. John's wort and sulfamethoxazol
* Galactosemia (lack of galactose-1-phosphat-uridylyltransferase or UDP-galactose-4-epimerase or galactokinase; Fanconi-Bickel-syndrome); congenital lack of lactase; glucose-galactose malabsorption
* Presence of one or more of the following eye disorders: cataract, retinopathia, optic neuropathy, alteration of the cornea
* Presence of one or more of the following laboratory abnormalities: anaemia, thrombocytopenia, leukopenia, neutropenia or agranulocytosis

Group A:

* Glucocorticoid naïve patients
* Start of glucocorticoid treatment or change in dosage <6 month prior to screening (dosing adaptations according to weight change are allowed)

Group B:

* Glucocorticoid treated patients or patients that stopped glucocorticoid treatment <6 month prior to screening
* Assisted ventilation of any kind necessary

Ages: 78 Months to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Reduction of disease progression | Baseline to week 48
  To test if tamoxifen treatment, compared to placebo, reduces the progression of the disease in 6.5-12 years old ambulant DMD patients (Group A) by at least 50% (using the MFM D1 subscore as primary clinical endpoint).

SECONDARY OUTCOMES:
Muscle function measured by D2 MFM subscore | Baseline to week 48
  D2 MFM subscore from baseline to week 48 under TAM treatment compared to placebo.
Muscle function measured by D3 MFM subscore | Baseline to week 48
  D3 MFM subscore from baseline to week 48 under TAM treatment compared to placebo.
Muscle function measured by North Star Ambulatory Assessment | Baseline to week 48
  North Star Ambulatory Assessment from baseline to week 48 under TAM treatment compared to placebo.
Muscle function measured by proximal upper limb function | Baseline to week 48
  Proximal upper limb function from baseline to week 48 under TAM treatment compared to placebo.
Muscle function measured by 6 minute walking distance in meter | Baseline to week 48
  6 minute walking distance in meter from baseline to week 48 under TAM treatment compared to placebo.
Muscle function measured by 10 meter walking time in seconds | Baseline to week 48
  10 meter walking time in seconds from baseline to week 48 under TAM treatment compared to placebo.
Muscle function measured by time to rise from lying on the floor / supine up in seconds | Baseline to week 48
  time to rise from lying on the floor / supine up in seconds from baseline to week 48 under TAM treatment compared to placebo.
Muscle force measured by quantitative muscle testing (using Myogrip) | Baseline to week 48
  Quantitative muscle testing (using Myogrip) from baseline to week 48 under TAM treatment compared to placebo.
Muscle Degeneration measured by MRI | Baseline to week 48
  Quantitative muscle MRI including muscle fat fraction (MFF) and T2 times of thigh muscles visualised by MRI from baseline to week 48 under TAM treatment compared to placebo.

OTHER OUTCOMES:
Patient reported outcome measured by PARS III questionnaire | Baseline to week 48
  Personal Adjustment and Role Skills Scale (PARS-III) from baseline to week 48 under TAM treatment under TAM treatment compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Fischer, MD, Principal Investigator — University Children's Hospital Basel
Locations (11):
- France (2):
  - Hôpitaux Raymond Poincaré, Garches
  - Hôpital de Hautepierre, Strasbourg
- Germany (2):
  - DRK Klinik Berlin Westend, Berlin
  - Universitätsklinikum Essen, Essen
- Radboud umc, Nijmegen, Netherlands
- Spain (2):
  - Hospital Sant Joan de Déu. UB, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
- University Children's Hospital Basel, Basel, Switzerland
- United Kingdom (3):
  - Royal Hospital for Children, Glasgow
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children's Hospital, Liverpool

REFERENCES:
- [Derived] Henzi BC, Putananickal N, Schmidt S, Nagy S, Rubino-Nacht D, Schaedelin S, Amthor H, Childs AM, Deconinck N, Horrocks I, Houwen-van Opstal S, Laugel V, Lobato ML, Osorio AN, Schara-Schmidt U, Spinty S, von Moers A, Lawrence F, Hafner P, Dorchies OM, Fischer D. Safety and efficacy of tamoxifen in non-ambulant patients with Duchenne muscular dystrophy: a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial (TAMDMD Group B). Neuromuscul Disord. 2025 Feb;47:105275. doi: 10.1016/j.nmd.2025.105275. Epub 2025 Jan 16. PMID 39879732
- [Derived] Henzi BC, Schmidt S, Nagy S, Rubino-Nacht D, Schaedelin S, Putananickal N, Stimpson G; North Star Consortium; Amthor H, Childs AM, Deconinck N, de Groot I, Horrocks I, Houwen-van Opstal S, Laugel V, Lopez Lobato M, Madruga Garrido M, Nascimento Osorio A, Schara-Schmidt U, Spinty S, von Moers A, Lawrence F, Hafner P, Dorchies OM, Fischer D. Safety and efficacy of tamoxifen in boys with Duchenne muscular dystrophy (TAMDMD): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2023 Oct;22(10):890-899. doi: 10.1016/S1474-4422(23)00285-5. PMID 37739572
- [Derived] Nagy S, Hafner P, Schmidt S, Rubino-Nacht D, Schadelin S, Bieri O, Fischer D. Tamoxifen in Duchenne muscular dystrophy (TAMDMD): study protocol for a multicenter, randomized, placebo-controlled, double-blind phase 3 trial. Trials. 2019 Nov 21;20(1):637. doi: 10.1186/s13063-019-3740-6. PMID 31752977